CLINICAL TRIAL: NCT06140888
Title: Effect of Ginkgo Biloba Extract on Cognitive Function in Acute Ischemic Stroke: a Multicentre, Randomised, Open-label, Blinded-Endpoint Trial
Brief Title: Effect of Ginkgo Biloba Extract on Cognitive Function in Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of the First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEFIT
Record Dates: First submitted 2023-11-15; First posted 2023-11-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ginkgo biloba extract group (Experimental): Ginkgo biloba extract 8 pills three times per day is administrated.
  Interventions: Drug: Ginkgo Biloba Extract
- The control group (No Intervention): Standard medical therapy

INTERVENTIONS:
Drug: Ginkgo Biloba Extract — Ginkgo biloba extract 8 pills three times per day is administrated.
  Arms: The ginkgo biloba extract group

SUMMARY:
The purpose of this study is to determine the effect of ginkgo biloba extract on cognitive function in acute ischemic stroke.

DETAILED DESCRIPTION:
Vascular brain injury is a common post-stroke complication that can reduce cognitive function and lead to vascular cognitive impairment, placing a significant burden on families and society. The purpose of this study is to determine the effect of ginkgo biloba extract on cognitive function in acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a definitive clinical diagnosis of acute ischemic stroke;
2. Age≥18 years, regardless of sex；
3. Primary education level or higher; baseline MoCA score of 10-25 points;
4. Able to complete cognitive scale scoring;
5. Informed consent is signed and ginkgo biloba extract therapy is initiated within 14 days of onset.

Exclusion Criteria:

1. Transient ischemic attack；
2. Patients who received emergency reperfusion therapy (including intravenous thrombolysis and endovascular thrombectomy) at onset;
3. Combined with other neurological diseases, such as neurodegenerative diseases (e.g., Alzheimer's disease, Parkinson's disease, Lewy body dementia, and frontotemporal dementia), optic neuritis, epilepsy, central nervous system infections (e.g., AIDS and syphilis), traumatic brain injury dementia, etc；
4. Currently using psychoactive medications (e.g., antidepressants) or anti-epileptic drugs, or if the time since their last use of these medications was less than 5 half-lives (per the pharmacokinetics of each specific medication; for drugs with unknown half-lives, a 1 month washout period was required)；
5. Had a pre-existing diagnosis of a cognitive disorder；
6. Currently taking medications intended to improve cognitive function or prevent dementia (e.g., cholinesterase inhibitors, memantine, nootropics), or if the washout period since their last use of these medications was less than 5 half-lives as specified in each drug's pharmacokinetics. For drugs with unknown half-lives, a minimum 1 month washout period was required；
7. Severe liver and kidney dysfunction;
8. Active ulcer or bleeding diathesis；
9. Allergy to preparations containing ginkgo biloba extract；
10. Pregnant or lactating women, patients with a life expectancy less than 6 months, and those unable to complete the study for other reason；
11. Unwillingness to be followed up or poor treatment compliance;
12. Those who are participating in other clinical investigators, or who have participated in other clinical studies within 3 months prior to enrollment;
13. Other conditions that the investigators deemed unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes of the Montreal Cognitive Assessment (MoCA) score | 180 days
  The MoCA scores in the 180 day of treatment minus baseline MoCA scores. MoCA scores range from 0 to 30, with higher MoCA scores indicating better cognitive function.

SECONDARY OUTCOMES:
Changes of the Mini-Metal State Examination (MMSE) score | 180 days
  The MMSE scores in the 180 day of treatment minus baseline MMSE scores. MMSE scores range from 0 to 30, with higher MMSE scores indicating better cognitive function.
the Montreal Cognitive Assessment (MoCA) score | 180 days
  MoCA scores range from 0 to 30, with higher MoCA scores indicating better cognitive function.
the Mini-Metal State Examination (MMSE) score | 180 days
  MMSE scores range from 0 to 30, with higher MMSE scores indicating better cognitive function.
the modified rankin scale (mRS) score | 90 days; 180 days
  mRS Scores range from 0 to 6, with a higher mRS Score indicating a worse prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, PhD, Principal Investigator — The First Hospital of Jilin University